CLINICAL TRIAL: NCT02648672
Title: A Single Ascending Dose Study to Examine the Safety, Tolerability, and Pharmacokinetic Profile of BPN14770 in Healthy Male and Female Subjects
Brief Title: BPN14770 Single Ascending Dose Study in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetra Discovery Partners (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPN14770-CNS-101
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — BPN14770

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BPN14770 (Experimental): A single oral dose of BPN14770.
  Interventions: Drug: BPN14770
- Placebo (Placebo Comparator): A single oral dose of placebo matching BPN14770
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BPN14770 — BPN14770 is an investigational new drug being developed for the treatment of Alzheimer's disease and other cognitive disorders. BPN14770 is a small molecule, subtype selective, negative allosteric modulator of phosphodiesterase 4D.
  Arms: BPN14770
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized double-blind (investigator and subject blinded), placebo controlled ascending single dose study to evaluate the safety, tolerability, and pharmacokinetic profile of BPN14770 in healthy male and female subjects. Each subject will be randomized to receive either a single dose of BPN14770 or placebo.

DETAILED DESCRIPTION:
Objectives:

1. To evaluate the safety and tolerability profile of single oral ascending dose levels of BPN14770 in healthy subjects.
2. To characterize the BPN14770 plasma pharmacokinetic profile following oral administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female. Female subjects must not be pregnant or breastfeeding.
2. Subject must be between 18 and 55 years of age (inclusive).
3. Subject's body mass index (BMI) must be between 18 and 32 kg/m2 (inclusive), and subject must weigh a minimum of 50 kg (110 lbs).
4. Female subjects must be surgically sterile (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 6 months prior to dosing) or at least 2 years postmenopausal. Menopausal status will be verified by a follicle-stimulating hormone (FSH) test at screening. In addition, all females must have a negative pregnancy test result within 48 hours before study drug administration regardless of childbearing potential.
5. Male subjects must be willing to inform female partners of their participation in the study and to use adequate contraceptive methods (must have had vasectomy at least 6 months prior to dosing or use at least one barrier method of birth control).
6. Subject must understand the study procedures, voluntarily consent to participate in this study, and provide their written informed consent prior to start of any study-specific procedures.
7. Subject is willing and able to remain in the study unit for the entire duration of the confinement period and return for outpatient visits.

Exclusion Criteria:

1. Clinically significant abnormality in the investigator's opinion indicated from the current hematology, biochemistry, or urinalysis tests, or from medical history, social history, vital signs, or physical examination.
2. Positive serology results for hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
3. Marked hypotension (systolic blood pressure [BP] ˂90 mmHg or diastolic BP ˂50 mmHg) or hypertension (systolic BP ˃160 mmHg or diastolic BP ˃100 mmHg) based on supine and sitting values at screening or predose. Out-of-range vital signs may be repeated once.
4. Marked bradycardia (heart rate ˂45 beats per minute [bpm]) or tachycardia (heart rate ˃110 bpm) based on supine, sitting, and ECG values at screening or predose. Out-of-range vital signs may be repeated once.
5. Current or past history of cardiovascular, cerebrovascular, pulmonary, renal, or liver disease.
6. History of hematological disorders (e.g., thrombocytopenia) in the immediate family (i.e, parents and siblings).
7. Clinically important or significant conduction abnormalities on average of triplicate ECGs (including QTc intervals ˃450 msec); evidence or history of long QT syndrome. This exclusion applies to the ECGs taken at screening, Day -1, and Day 1 predose.
8. Current or past history of gastric or duodenal ulcers or other diseases of the gastrointestinal tract that could interfere with absorption of study drug. Note: Subject with history of appendectomy or cholecystectomy may be enrolled.
9. Active acute or chronic infectious diseases.
10. Unable to discontinue any over the counter (OTC) medication utilized on a regular basis or has taken any prescription medication within 14 days prior to admission to the study on Day -2.
11. Regular (daily) consumption of alcohol exceeding two servings of beer or the equivalent amount of other forms of alcohol (1 serving = 12 oz beer, 5.0 oz wine, or 1.5 oz distilled spirits).
12. Any history of alcohol or drug abuse within the previous year prior to the Screening Visit (per the current edition of the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition: DSM-5).
13. Any use of alcohol within 48 hours of admission into the study on Day -2.
14. Active smokers or tobacco users (e.g., chew and snuff) who are unable to discontinue tobacco use at least 6 months prior to admission to the study on Day -2 and refrain from using tobacco during the study treatment and evaluation period.
15. Inability or unwillingness to comply with the protocol or rules of the clinical research unit, or likely inability to complete the study.
16. Participation in other clinical studies involving investigational drug within the previous 30 days prior to the Screening Visit.
17. Donation of blood or blood products (including plasma) during the 8 weeks before the first administration of study drug on Day 1.
18. Positive screen for drugs of abuse.
19. History of allergy to penicillin or sulfonamides, or any other clinically significant drug allergy that includes symptoms such as shortness of breath, rash, or edema.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1 week
  Incidence and nature of adverse events (AEs) and serious adverse events (SAEs). Significant assessments reported as AEs or SAEs include clinical laboratory assessments and vital signs, physical and neurological examination, 12-lead electrocardiogram (ECG)

SECONDARY OUTCOMES:
Area Under the Curve from Time Zero Extrapolated to Infinity [AUC0-∞] | 48 hr
Maximum Concentration [Cmax] | 48 hr

CONTACTS AND LOCATIONS:
Overall Officials: Scott Reines, MD, PhD, Study Chair — Tetra Discovery Partners
Locations (1):
- Jasper Clinic, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No